CLINICAL TRIAL: NCT05746598
Title: Effect of Genetic and Epigenetic Factors on the Clinical Response and Toxicity to Cisplatin Among Egyptian Non-small Cell Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer, Misr International University
Other Study IDs: NSCLC-Genetics
Record Dates: First submitted 2023-02-08; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Non Small Cell Lung Cancer; Nephropathy; Cardiotoxicity
Keywords: Non-small cell lung Cancer; Nephropathy; Cardiotoxicity; Gene polymorphism; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Kidney Diseases; Cardiotoxicity | interventions — Cisplatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: NSCLC patients Who developed Toxicity to Chemotherapeutic agents
  Interventions: Drug: Cisplatin injection
- 2: NSCLC patients Who did not developToxicity to Chemotherapeutic agents
  Interventions: Drug: Cisplatin injection

INTERVENTIONS:
Drug: Cisplatin injection — Cisplatin 75mg/m2

SUMMARY:
Lung cancer is the leading cause of death worldwide, with non-small-cell lung cancer (NSCLC) being the most common histotype according to the global cancer observatory 2022. A variety of therapeutic options for advanced/metastatic non-oncogene-addicted NSCLC have recently been approved based on their impact on patient outcomes in terms of survival and safety profile. Current guidelines advocate for personalized treatment options based on molecular and immunologic characteristics, which drives the physician's decision toward tailored oncology.

In the last two to three decades, hundreds of cancer biological prognostic markers for non-small cell lung cancer have been proposed. Although they have shown a potential in this ﬁeld, validation studies are still required and, to date, there is in suﬃcient evidence to recommend the routine clinical use of any of these putative biomarkers. Therefore, the discovery of robust prognostic and/or predictive biomarkers in patients with non-small cell lung cancer is imperative for advancing treatment strategies for the disease and improving patient care.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC cancer patients treated with Cisplatin-containing chemotherapy.
* Measurable disease.
* Age of 18 years to 80 years.

Exclusion Criteria:

* Non-small cell lung cancer patients who had undergone radiotherapy or chemotherapy.
* Pregnant and lactating females.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin.
* Any other medical or psychiatric condition or severe or chronic laboratory abnormality making the inclusion of the patient in the study inappropriate in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • NSCLC cancer patients treated with Cisplatin-containing chemotherapy.
Sampling Method: Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Nephrotoxicity | 6 months
  Change in Creatinine Clearance

SECONDARY OUTCOMES:
Blood urea nitrogen | 6 months
  Change in Blood urea nitrogen
Serum creatinine | 6 month
  change in Serum creatinine
Cardiotoxicity | 6 months
  Change in ejection fraction

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided